CLINICAL TRIAL: NCT01376297
Title: A Phase III, Multicenter, Randomized, Double-blind, Unbalanced (3:1) Active Control Study to Assess the Safety and Describe the Efficacy of Netupitant and Palonosetron for the Prevention of Chemotherapy-induced Nausea and Vomiting in Repeated Chemotherapy Cycles.
Brief Title: A Safety Study of Oral Netupitant and Palonosetron for the Prevention of Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NETU-10-29
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — netupitant, palosentron drug combination; Aprepitant; Palonosetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Netupitant and Palonosetron plus dexamethasone (Experimental): Oral netupitant/palonosetron (300 mg/0.50 mg) hard capsule (on Day 1) with oral dexamethasone prior to each scheduled chemotherapy cycle
  Interventions: Drug: Netupitant and Palonosetron; Drug: Dexamethasone
- Aprepitant and Palonosetron plus dexamethasone (Active Comparator): Oral aprepitant hard capsule 125 mg (on Day 1) + 80 mg daily (for the following two days) and oral palonosetron soft capsule 0.50 mg (on Day 1) given with oral dexamethasone at each scheduled chemotherapy cycle.
  Interventions: Drug: Aprepitant; Drug: Palonosetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Netupitant and Palonosetron
  Arms: Netupitant and Palonosetron plus dexamethasone
Drug: Aprepitant
  Arms: Aprepitant and Palonosetron plus dexamethasone
Drug: Palonosetron
  Arms: Aprepitant and Palonosetron plus dexamethasone
Drug: Dexamethasone

SUMMARY:
NETU-10-29 is a clinical study assessing safety of netupitant and palonosetron, two antiemetic drugs, both given with oral dexamethasone. The objective of the study is to evaluate if netupitant and palonosetron are safe when administered to prevent nausea and vomiting after administration of repeated cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Naïve to cytotoxic chemotherapy. Previous biological or hormonal therapy is permitted.
* Diagnosed with a malignant tumor.
* If scheduled to receive repeated consecutive courses of chemotherapy, a single dose of one or more of the following agents administered on Day 1 is allowed:

  * Highly emetogenic chemotherapy: any I.V. dose of cisplatin, mechlorethamine, streptozocin, cyclophosphamide more or equal to 1500 mg/m2, carmustine, dacarbazine;
  * Moderately emetogenic chemotherapy: any I.V. dose of oxaliplatin, carboplatin, epirubicin, idarubicin, ifosfamide, irinotecan, daunorubicin, doxorubicin, cyclophosphamide I.V. (less than 1500 mg/m2), cytarabine I.V. (more than 1 g/m2), azacidine, alemtuzumab, bendamustine, or clofarabine.
* If scheduled to receive combination regimens, the most emetogenic agent is to be given as first on Day 1 and the infusion must be completed within 6 hours.
* If scheduled to receive chemotherapy agents of minimal to low emetogenic potential, they are to be given on Day 1 following the most emetogenic agent or on any subsequent study day.
* ECOG Performance Status of 0, 1, or 2
* Female patients of either non-childbearing potential or child-bearing potential with a commitment to use contraceptive methods throughout the clinical trial
* Hematologic and metabolic status adequate for receiving a moderately emetogenic regimen based on laboratory criteria (Total Neutrophils,Platelets, Bilirubin, Liver enzymes, Serum Creatinine or Creatinine Clearance)

Exclusion Criteria:

* If female, lactating or pregnant
* Current use of illicit drugs or current evidence of alcohol abuse.
* Scheduled to receive either cyclophosphamide I.V. (500 to 1500 mg/m2) and I.V. doxorubicin (more or equal to 40 mg/m2) or cyclophosphamide I.V. (500 to 1500 mg/m2) and I.V. epirubicin (more or equal to 60 mg/m2).
* Scheduled to receive moderately or highly emetogenic chemotherapy from Day 2 to Day 5 following Day 1 chemotherapy administration.
* Active infection or uncontrolled disease except for malignancy that may pose unwarranted risks in administering the study drugs to the patient.
* Known hypersensitivity or contraindication to 5-HT3 receptor antagonists or dexamethasone.
* Previously received an NK1 receptor antagonist
* Participation in a clinical trial involving oral netupitant administered in combination with palonosetron.
* Any investigational drugs taken within 4 weeks prior to Day 1 of cycle 1, and/or is scheduled to receive any investigational drug during the study.
* Systemic corticosteroid therapy at any dose within 72 hours prior to Day 1 of cycle 1. Topical and inhaled corticosteroids with a steroid dose of less or equal to 10 mg of prednisone daily or its equivalent are permitted. Non-study drug dexamethasone as pre-medication in patients scheduled to receive taxanes is allowed.
* Scheduled to receive bone marrow transplantation and/or stem cell rescue therapy.
* Scheduled to receive any strong or moderate inhibitor of CYP3A4 or its intake within 1 week prior to Day 1
* Scheduled to receive any of the following CYP3A4 substrates: terfenadine, cisapride, astemizole, pimozide.
* Scheduled to receive any CYP3A4 inducer or its intake within 4 weeks prior to Day 1
* History or predisposition to cardiac conduction abnormalities, except for incomplete right bundle branch block.
* History of risk factors for Torsade de Point (heart failure, hypokalemia, family history of Long QT Syndrome).
* Severe cardiovascular diseases within 3 months prior to Day 1, including myocardial infarction, unstable angina pectoris, significant valvular or pericardial disease, history of ventricular tachycardia, symptomatic Congestive Heart Failure and severe uncontrolled arterial hypertension.
* Any illness or condition that, in the opinion of the investigator, may confound the results of the study or pose unwarranted risks in administering the investigational product to the patient.
* Concurrent medical condition that would preclude administration of dexamethasone for 4 days such as systemic fungal infection or uncontrolled diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (75):
- United States (11):
  - Northwest Alabama Cancer Center PC, Muscle Shoals, Alabama
  - East Valley Hematology and Oncology Medical Group, Burbank, California
  - American Institute of Research, Los Angeles, California
  - Veterans Administration New Jersey Health Care System, East Orange, New Jersey
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Hematology and Oncology Associates, Inc., Canton, Ohio
  - Tri-County Hematology & Oncology Associates, Inc, Massillon, Ohio
  - Cancer Center at Memorial Hospital of RI, Pawtucket, Rhode Island
  - Spartanburg Regional Health Services, Spartanburg, South Carolina
  - South Texas Comrehensive Cancer Centers, Corpus Christi, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Bulgaria (5):
  - UMHAT "Dr. Georgi Stranski", Pleven
  - Complex Oncology Center - Shumen Ltd. [Oncology], Shumen
  - Specialized Hospital for Active Treatment in Oncology "Dr. Marko Markov" Varna, Varna
  - COC - Veliko Tarnovo Dept. Medical Oncology, Veliko Tarnovo
  - COC - Vratsa Dept. of Palliative Care, Vratsa
- Czechia (5):
  - Oblastni nemocnice Mlada Boleslav a.s., Onkologie, Mladá Boleslav
  - AVICENNUS s.r.o. Onkologie Nymburk, Nymburk
  - Fakultni nemocnice v Motole, Prague
  - Nemocnice Na Homolce, Oddeleni klinicke onkologie, Prague
  - Nemocnice Znojmo, p.o., Znojmo
- Germany (11):
  - Gemeinschaftspraxis, Dr. Med O.Brundler und B.Heinreich, PD Dr. med M.Bangerter Fachärzte für Innere Medizin, Hämatologie und internistische Onkologie, Augsburg
  - Charite - Campus Benjamin Franklin (CBF), Berlin
  - Medizinisches Versorgungszentrum für Hämatologie und Tumorerkrankungen, HIV/AIDS und Hepatitiden, Berlin
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - St. Johannes Hospital Medizinische Klinik II, Hämatologie, Onkologie und klinische Immunologie, Duisburg
  - Praxis Fuer Interdisziplinaere Onkologie und Haematologie, Freiburg im Breisgau
  - Medizinische Hochschule, Zentrum für Innere Medizin, Klinik für Hämatologie, Hämostaseologie, Onkologie und Stammzelltransplantation, Hanover
  - Ärzteforum Hennigsdorf, Hennigsdorf
  - Praxis für Innere Medizin, Hämatologie und Internistische Onkologie, Marburg
  - Krankenhaus, Maria Hilf, St. Franziskus Innere Medizin, Mönchengladbach
  - OncoPRO GbR Dr. R. Dengler, Dr. A. Kröber, Regensburg
- Hungary (6):
  - Országos Onkológiai Intézet, B. Belgyógyászati Osztály, Budapest
  - Bekes Megyei Kepviselo-testulet Pandy Kalman Korhaz, Gyula
  - Kaposi Mor Oktato Korhaz [Klinikai Onkologiai Centrum], Kaposvár
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktatók, Miskolc
  - Dr. Bugyi Istvan Korhaz [Oncology], Szentes
  - Fejér Megyei Szent György Kórház [Onkológiai Osztály], Székesfehérvár
- India (9):
  - Kumaran Hospital PVT Ltd, Chennai
  - Dr.Rai Memorial Medical centre, Chennai
  - Acharya Harihara Regional Cancer Centre [Oncology], Cuttack
  - M.S Patel Cancer Hospital [Oncology], Gujarat
  - Research Unit, The Karnatak cancer therapy & Research Instit, Hubli
  - S.M.S College And Hospital, Jaipur
  - Apollo Speciality Hospital [Oncology], Madurai
  - Lucknow Cancer Institute [Oncology], Uttar Pradesh
  - King George Hospital [Medical Oncology], Visakhapatnam
- Poland (7):
  - Bialostockie Centrum Onkologii im. M.Sklodowskiej-Curie im dr. E.Pileckiej z Pododdzialem Chemioterapii Dziennej, Bialystok
  - Centrum Onkologii Ziemi Lubelskiej im.Sw.Jana z Dukli III Oddzial Onkologii Ginekologicznej, Radioterapii I Chemioterapii, Lublin
  - Ginekologiczno-Położniczy Szpital Kliniczny UM w Poznaniu, Poznan
  - Szpital Kliniczny Przemienienia Panskiego UM w Poznaniu, Poznan
  - Wielkopolskie Centrum Onkologii im. M. Sklodowskiej-Curie i Onkologii Ginekologicznej, Poznan
  - Szpital Specjalistyczny, Prabuty
  - Szpital Rejonowy im. dr J. Rostka w Raciborzu, Racibórz
- Russia (10):
  - GBUZ "Cheliabinsky Regional Oncology Dispensary", Chelyabinsk
  - GAUZ Republican Clinical Oncology Dispensary of Minzdrav of Republic of Tatarstan, Kazan'
  - Non-State healthcare Indtitution Central Clinical Hospital # 2 named after N.A. Semashko OAO "RZhD", Moscow
  - Regional GUZ Orlovskiy Oncological Dispensary, Oryol
  - GUZ Leningradskiy Regional Oncology Dispensary, Saint Petersburg
  - GBOU VPO "Saint-Petersburg State Medical University, Saint Petersburg
  - GUZ Tula Regional Oncological Dispensary [Oncology], Tula
  - GBUZ Tyumen Regional Oncology Dispensary, Tyumen
  - GBUZ Republican Clinical Oncology Dispensary of Minzdrav of Republic of Bashkortostan, Ufa
  - FBUZ Privolzhsky District Medical Center of FMBA, Veliky Novgorod
- Serbia (3):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Institute of oncology and radiology of Serbia, Belgrade
  - Clinical Center Kragujevac, Kragujevac
- Ukraine (8):
  - Chernivtsi Regional Cancer Hospital [Outpatient Department], Chernivtsi
  - Komunalnyi zaklad Miska bahatoprofilna klinichna likarnia #4, Dnipropetrovks
  - KZ MKL19, MOTsr, vd khimter [viddilennia khimioterapii], Dnipropetrovsk
  - KKLPZ DnOPTsr [radio vd#3], Donetsk
  - DU IMR AMNU [vd khemter], Kharkiv
  - Poltavskyi oblasnyi klinichnyi onkolohichnyi dyspanser Pol, Poltava
  - Zakarpatskyi oblasnyi klinichnyi onkodyspanser [viddilennia, Uzhhorod
  - ZaOKOD [abdom vd], Zaporizhia

REFERENCES:
- [Derived] Schwartzberg L, Karthaus M, Rossi G, Rizzi G, Borroni ME, Rugo HS, Jordan K, Hansen V. Fixed combination of oral NEPA (netupitant-palonosetron) for the prevention of acute and delayed chemotherapy-induced nausea and vomiting in patients receiving multiple cycles of chemotherapy: Efficacy data from 2 randomized, double-blind phase III studies. Cancer Med. 2019 May;8(5):2064-2073. doi: 10.1002/cam4.2091. Epub 2019 Apr 9. PMID 30968588
- [Derived] Rugo HS, Rossi G, Rizzi G, Aapro M. Efficacy of NEPA (netupitant/palonosetron) across multiple cycles of chemotherapy in breast cancer patients: A subanalysis from two phase III trials. Breast. 2017 Jun;33:76-82. doi: 10.1016/j.breast.2017.02.017. Epub 2017 Mar 10. PMID 28285236

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 413 patients were randomized (ITT population), 412 patients received study drugs i.e.netupitant/palonosetron combination or aprepitant/palonosetron regimen, both with dexamethasone (safety population)
Groups:
- Netupitant and Palonosetron Plus Dexamethasone: Oral netupitant/palonosetron (300 mg/0.50 mg) hard capsule (on Day 1) with oral dexamethasone prior to each scheduled chemotherapy cycle
  Netupitant and Palonosetron
  Dexamethasone
- Aprepitant and Palonosetron Plus Dexamethasone: Oral aprepitant hard capsule 125 mg (on Day 1) + 80 mg daily (for the following two days) and oral palonosetron soft capsule 0.50 mg (on Day 1) given with oral dexamethasone at each scheduled chemotherapy cycle.
  Aprepitant
  Palonosetron
  Dexamethasone
Period: Overall Study
Arm/Group | Netupitant and Palonosetron Plus Dexamethasone | Aprepitant and Palonosetron Plus Dexamethasone
Started | 309 (number of randomised patients) | 104 (number of randomised patients)
Completed | 181 (number of patients completing planned/unplanned chemotherapy cycles) | 55 (number of patients completing planned/unplanned chemotherapy cycles)
Not Completed | 128 | 49

BASELINE CHARACTERISTICS:
Population: Safety Population, i.e. patients receiving study drugs (either netupitant/palonosetron combination or aprepitant/palonosetron regimen, both with dexamethasone)
Groups:
- Total: Total of all reporting groups
Arm/Group | Netupitant and Palonosetron Plus Dexamethasone | Aprepitant and Palonosetron Plus Dexamethasone | Total
Number analyzed (Participants) | 308 | 104 | 412
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.44) | 56.9 (11.70) | 56.6 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 51 | 206
  Male | 153 | 53 | 206
Race/Ethnicity, Customized [Number; unit: participants]
  White | 258 | 87 | 345
  Black | 3 | 0 | 3
  Asian | 47 | 17 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Adverse Events
Description: This was a safety study where Adverse Events is the primary outcome (defined by the current ICH Guideline for Good Clinical Practice). Patients were randomized according to a 3:1 ratio (netupitant/palonosetron:aprepitant/palonosetron). No formal comparison was planned, the presence of a control in the same patient population helped interpret any unexpected safety finding in the experimental arm.The number of patients was estimated in order to have more than 100 patients treated with the netupitant/palonosetron comination for up to at least six cycles. Based on 100 patients, if a given AE is not observed, an AE incidence of 3% or greater can be excluded with 95% confidence.
Time Frame: Participants will be followed for the duration of the chemotherapy, an expected average duration of up to 24 weeks assuming 6 chemotherapy cycles given every 4 weeks
Population: Safety Population
Measure: Number; unit: percentage of patients with TEAE
Arm/Group | Netupitant and Palonosetron Plus Dexamethasone | Aprepitant and Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 308 | 104
percentage of patients with TEAE | 86.0 | 91.3

ADVERSE EVENTS:
Time Frame: The reporting period for AEs was the period starting from the time of informed consent signature until 21 (+2) days post study drug administration (Day 1 of last cycle).
Description: Based on the medical judgment of the investigator, all non resolved, non serious AEs beyond this date could have been followed for an additional 14 days. At the end of this additional follow up period, all unresolved AEs were documented on the eCRF as 'ongoing.'
Arm/Group | Netupitant and Palonosetron Plus Dexamethasone | Aprepitant and Palonosetron Plus Dexamethasone
Serious Adverse Events (participants affected / at risk) | 50/308 | 19/104
Other Adverse Events (participants affected / at risk) | 265/308 | 95/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Netupitant and Palonosetron Plus Dexamethasone (N=308) | Aprepitant and Palonosetron Plus Dexamethasone (N=104)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 3 | 0
Long QT syndrome (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1
Asthenia (General disorders) | 2 | 0
Device dislocation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chemotherapy extravasation management (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Netupitant and Palonosetron Plus Dexamethasone (N=308) | Aprepitant and Palonosetron Plus Dexamethasone (N=104)
Anaemia (Blood and lymphatic system disorders) | 58 | 26
Leukopenia (Blood and lymphatic system disorders) | 55 | 18
Neutropenia (Blood and lymphatic system disorders) | 95 | 29
Thrombocytopenia (Blood and lymphatic system disorders) | 38 | 16
Constipation (Gastrointestinal disorders) | 26 | 9
Diarrhoea (Gastrointestinal disorders) | 32 | 19
Dyspepsia (Gastrointestinal disorders) | 16 | 3
Nausea (Gastrointestinal disorders) | 18 | 11
Stomatitis (Gastrointestinal disorders) | 9 | 6
Asthenia (General disorders) | 30 | 12
Fatigue (General disorders) | 29 | 15
Pyrexia (General disorders) | 19 | 10
Blood creatinine increased (Investigations) | 6 | 6
Neutrophil count decreased (Investigations) | 17 | 4
Decreased appetite (Metabolism and nutrition disorders) | 20 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 16 | 4
Headache (Nervous system disorders) | 15 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 77 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor and investigator(s) agree that no publications discussing trials' results will occur until release of final report. Sponsor has no objections if the investigators publish study results, however the investigator is requested to contact the sponsor before publishing, to prevent premature disclosure of data and is not intended as a restrictive measure concerning results or opinions of investigators.